CLINICAL TRIAL: NCT01836471
Title: A Double-blind, Placebo-controlled, Study Examining the Effect of Orally Administered QAW039 (450 mg QD) on FEV1 and ACQ in Non-atopic, Asthmatic Patients With a Baseline, Pre-bronchodilator FEV1 of 40-80% Predicted, Inadequately Controlled With Low Dose ICS Therapy
Brief Title: A Study to Assess the Effect of QAW039 in Non-atopic Asthmatic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAW039A2214; 2012-003995-38 (EudraCT Number)
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — fevipiprant; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- QAW039 450 mg qd Non-atopic (Experimental): QAW039 450 mg (3 capsules of QAW039 150 mg) qd combined with background ICS (100 μg fluticasone, bid). Non-atopic patients randomized in ratio of approximately 1:1.
  Interventions: Drug: QAW039; Drug: Fluticasone 100 mcg
- Placebo Non-atopic (Placebo Comparator): Placebo to QAW039 (3 capsules of Placebo of QAW039 150 mg) combined with background ICS (100 μg fluticasone, bid). Non-atopic randomized in ratio of approximately 1:1.
  Interventions: Drug: Placebo QAW039; Drug: Fluticasone 100 mcg
- QAW039 450 mg qd Atopic (Experimental): QAW039 450 mg (3 capsules of QAW039 150 mg) qd combined with background ICS (100 μg fluticasone, bid). Atopic patients randomized in a ratio of approximate 1:1:1
  Interventions: Drug: QAW039; Drug: Fluticasone 100 mcg
- Fluticasone 150 mcg bid Atopic (Active Comparator): Placebo to QAW039 (3 capsules of Placebo of QAW039 150 mg) combined with 150 μg ICS and with background ICS (100 μg fluticasone, bid). As a consequence total ICS was 250 μg fluticasone bid. Atopic patients randomized in ratio of approximately 1:1:1
  Interventions: Drug: Placebo QAW039; Drug: Fluticasone 250 mcg
- Placebo Atopic (Placebo Comparator): Placebo to QAW039 (3 capsules of Placebo of QAW039 150 mg) combined with background ICS (100 μg fluticasone, bid). Atopic patients andomized in ratio of approximately 1:1:1
  Interventions: Drug: Placebo QAW039; Drug: Fluticasone 100 mcg

INTERVENTIONS:
Drug: QAW039 — QAW039 supplied as hard gelatin capsule in unit dose strength of 150 mg. Patient took 450 mg once daily (3 capsules taken with food in the morning) for the approximate period of the study (12 weeks)
  Arms: QAW039 450 mg qd Atopic; QAW039 450 mg qd Non-atopic
Drug: Placebo QAW039 — Matching placebo for QAW039 supplied as hard gelatin capsule were identical in appearance to their active counterparts. Patients took 3 QAW039 matching placebo capsules once a day ( taken with food in the morning) for the approximate period of the study (12 weeks)
  Arms: Fluticasone 150 mcg bid Atopic; Placebo Atopic; Placebo Non-atopic
Drug: Fluticasone 250 mcg — Fluticasone was supplied in inhalers with dose strength of 250 mcg. Patients took 250 mcg bid (morning and evening approximately 12 hours between doses) for a total dose of 500 mcg daily for the approximate period of the study (12 weeks).
  Arms: Fluticasone 150 mcg bid Atopic
Drug: Fluticasone 100 mcg — Background therapy - fluticasone was supplied in inhalers with dose strength of 100 mcg. All patients in the study other than the Atopic Fluticasone 150 mcg arm were given the 100 mcg dose strength inhalers and took fluticasone 100 mcg bid (taken morning and evening with approximately 12 hours between doses) as background therapy for the approximate period of the study (12 weeks).
  Arms: Placebo Atopic; Placebo Non-atopic; QAW039 450 mg qd Atopic; QAW039 450 mg qd Non-atopic

SUMMARY:
The purpose of the study was to assess the clinical effect of QAW039 in non-atopic asthmatics taking low dose Inhaled Corticosteroid (ICS) as background therapy.

DETAILED DESCRIPTION:
This was a multi-centre, randomised, placebo-controlled, double blind, 3-arm study designed to compare the efficacy and safety of a once daily dose of QAW039 with placebo in non-atopic and atopic asthmatics both inadequately controlled despite receiving a low dose ICS background therapy, over a 12 week treatment period. Efficacy and safety of a once daily dose of QAW039 was also compared with an increased dose of ICS in atopic asthmatics taking low dose ICS as background therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed
* Patients with a diagnosis of persistent asthma (according to Global Initiative for Asthma 2011) for a period of at least 6 months prior to screening
* Patients with a pre-bronchodilator Forced Expiratory Volume In One Second (FEV1) value of 40% to 80% of individual predicted value at screening and prior to treatment
* An Asthma Control Questionnaire score ≥ 1.5 prior to treatment
* Demonstration of reversible airway obstruction

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Acute illness other than asthma at the start of the study
* Patients with clinically significant laboratory abnormalities at screening
* Patients with clinically significant condition which may compromise subject safety or interfere with study evaluation
* Use of other investigational drugs at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2013-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kay, Study Director — Novartis Pharmaceuticals
Locations (67):
- United States (27):
  - Novartis Investigative Site, Encinitas, California
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Mission Viejo, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Palmdale, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, Rolling Hills Estates, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Jose, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Papillion, Nebraska
  - Novartis Investigative Site, Skillman, New Jersey
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Lincoln, Rhode Island
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Seattle, Washington
- Belgium (2):
  - Novartis Investigative Site, Erpent
  - Novartis Investigative Site, Liège
- Colombia (4):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bogotá, Cundinamarca
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Medellín
- Czechia (4):
  - Novartis Investigative Site, Trutnov, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Karlovy Vary-Stara Rokle, CZE
  - Novartis Investigative Site, Teplice, CZE
- Germany (7):
  - Novartis Investigative Site, Marburg, Germany
  - Novartis Investigative Site, Wiesbaden, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Witten
- India (4):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Panjim, Goa
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
- Poland (3):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Wroclaw
- Romania (7):
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Bucharest, District 3
  - Novartis Investigative Site, Craiova, Dolj
  - Novartis Investigative Site, Timișoara, Romania
  - Novartis Investigative Site, Arad
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Deva
- South Africa (4):
  - Novartis Investigative Site, Durban, South Africa
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Gatesville
  - Novartis Investigative Site, Pretoria
- South Korea (5):
  - Novartis Investigative Site, Gwangju, Gwangju
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Cheongju-si, North Chungcheong

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 939 subjects were screened, 679 entered the inhaled corticosteroid (ICS) tapering run-in, 345 subjects were randomized; eleven randomized subjects discontinued the study prior to start of study drug. Patient disposition and baseline characteristics were presented for 334 subjects (received study drug)
Groups:
- QAW039 450 mg qd Non-atopic: QAW039 450 mg qd plus background ICS (100 μg fluticasone, bid). Non-atopic patients randomized in ratio of approximately 1:1 to QAW039 or placebo.
- Placebo Non-atopic: Placebo to QAW039 450 mg qd plus background ICS (100 μg fluticasone, bid). Non-atopic patients randomized in ratio of approximately 1:1 to QAW039 or placebo.
- QAW039 450 mg qd Atopic: QAW039 450 mg qd plus background ICS (100 μg fluticasone, bid). Atopic patients randomized in ratio of approximately 1:1:1 to QAW039 or fluticasone or placebo.
- Fluticasone 150 µg Bid Atopic: Fluticasone 150 µg plus background ICS (100 μg fluticasone, bid). Atopic patients randomized in ratio of approximately 1:1:1 to QAW039 or fluticasone or placebo.
- Placebo Atopic: Placebo to QAW039 450 mg qd plus background ICS (100 μg fluticasone, bid). Atopic patients randomized in ratio of approximately 1:1:1 to QAW039 or fluticasone or placebo.
Period: Overall Study
Arm/Group | QAW039 450 mg qd Non-atopic | Placebo Non-atopic | QAW039 450 mg qd Atopic | Fluticasone 150 µg Bid Atopic | Placebo Atopic
Started | 93 | 94 | 51 | 42 | 54
Completed | 82 | 85 | 49 | 40 | 49
Not Completed | 11 | 9 | 2 | 2 | 5
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 1 | 0 | 2
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 6 | 3 | 1 | 1 | 2
Not completed — Non compliance with tx | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QAW039 450 mg qd Non-atopic | Placebo Non-atopic | QAW039 450 mg qd Atopic | Fluticasone 150 µg Bid Atopic | Placebo Atopic | Total
Number analyzed (Participants) | 93 | 94 | 51 | 42 | 54 | 334
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (14.33) | 53.5 (14.37) | 50.3 (12.75) | 48.2 (12.16) | 48.2 (13.58) | 51.0 (13.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 26 | 23 | 25 | 194
  Male | 33 | 34 | 25 | 19 | 29 | 140
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 3 | 3 | 3 | 2 | 13
  Asian | 15 | 16 | 4 | 6 | 3 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 6 | 6 | 3 | 3 | 4 | 22
  White | 68 | 68 | 40 | 29 | 43 | 248
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
  Other | 2 | 1 | 1 | 1 | 1 | 6
Duration of asthma [Mean (Standard Deviation); unit: years] | 14.88 (12.349) | 12.82 (12.196) | 24.69 (17.446) | 27.78 (18.039) | 24.09 (16.055) | 18.91 (15.648)
Subject population [Number; unit: Participants] — Non-atopic defined as history of perennial symptoms with no clear inhaled allergic trigger AND a negative skin prick test (< 3mm diameter above background) or a negative specific IgE (<0.35 IU eq./ml). Atopic/allergic defined as skin prick test (≥ 3mm diameter above background) or a positive specific IgE (e.g.,RAST/CAP) test (≥0.35 IU eq/ml)
  Participants
    Non-atopic | 93 | 94 | 0 | 0 | 0 | 187
    Atopic | 0 | 0 | 51 | 42 | 54 | 147
Percentage of predicted FEV1 (%) pre-bronchodilator [Mean (Standard Deviation); unit: Percentage] | 67.5446 (11.81404) | 65.7286 (13.94056) | 69.0662 (12.16292) | 68.7483 (10.52156) | 64.8709 (12.97729) | 66.9849 (12.56166)
ACQ-6 score [Mean (Standard Deviation); unit: points] — Number of participants (n=92,94,51,42,54)
  points | 1.70 (0.762) | 1.53 (0.745) | 1.55 (0.665) | 1.68 (0.749) | 1.72 (0.675) | 1.63 (0.728)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough FEV1 (L) in Non-atopic Patients at Week 12 - Full Analysis Set
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Baseline is defined as the last available FEV1 measurement taken prior to the first dose of randomized study drug.
  Data within 6 hr of rescue medication use is excluded from this analysis. For subjects with missing trough FEV1 (L) at Week 12, the last post baseline observation were used (LOCF).
  Estimates are from a mixed effects model with treatment, subject population (non-atopic vs. atopic), treatment by subject population interaction, baseline trough FEV1 and region as fixed effects and center nested within region as random effects. Full analysis set included all randomized subjects who received at least one dose of study drug.
Time Frame: baseline,12 weeks
Measure: Least Squares Mean (Standard Error); unit: liter
Arm/Group | QAW039 450 mg qd Non-atopic | Placebo Non-atopic
Number analyzed (Participants) | 91 | 93
liter | 0.05 (0.029) | 0.03 (0.029)
Statistical Analysis 1: Comparison: QAW039 450 mg qd Non-atopic vs Placebo Non-atopic; Test type: Superiority or Other; p = 0.7269, Mixed Models Analysis; least squares mean = 0.01, 90% CI 2-sided [-0.5 to 0.08], Standard Error of Mean 0.038

2. Secondary Outcome: Change From Baseline in Trough FEV1 (L) in Atopic Patients at Week 12 - Full Analysis Set
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Baseline is defined as the FEV1 measurement taken prior to the first dose of randomized study drug.
  Data within 6 hr of rescue medication use is excluded from this analysis. For subjects with missing trough FEV1 (L) at Week 12, the last post baseline observation were used (LOCF).
  Estimates are from a mixed effects model with treatment, subject population (non-atopic vs. atopic), treatment by subject population interaction, baseline trough FEV1 and region as fixed effects and center nested within region as random effects. Full analysis set included all randomized subjects who received at least one dose of study drug.
Time Frame: baseline,12 weeks
Measure: Least Squares Mean (Standard Error); unit: liter
Arm/Group | QAW039 450 mg qd Atopic | Fluticasone 150 µg Bid Atopic | Placebo Atopic
Number analyzed (Participants) | 50 | 41 | 52
liter | 0.06 (0.038) | 0.01 (0.042) | 0.05 (0.037)
Statistical Analysis 1: Comparison: QAW039 450 mg qd Atopic vs Placebo Atopic; Test type: Superiority or Other; least sqares mean = 0.01, 90% CI 2-sided [-0.08 to 0.09], Standard Error of Mean 0.050
Statistical Analysis 2: Comparison: QAW039 450 mg qd Atopic vs Fluticasone 150 µg Bid Atopic; Test type: Superiority or Other; least squares mean = 0.04, 90% CI 2-sided [-0.04 to 0.13], Standard Error of Mean 0.054
Statistical Analysis 3: Comparison: Fluticasone 150 µg Bid Atopic vs Placebo Atopic; Test type: Superiority or Other; least squares mean = -0.04, 90% CI 2-sided [-0.13 to 0.05], Standard Error of Mean 0.053

3. Secondary Outcome: Change From Baseline in Trough FEV1 (L) in Non-atopic Compared to Atopic Patients at Week 12 - Full Analysis Set
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Baseline is defined as the FEV1 measurement taken prior to the first dose of randomized study drug.
  Data within 6 hr of rescue medication use is excluded from this analysis. For subjects with missing trough FEV1 (L) at Week 12, the last post baseline observation were used (LOCF).
  Estimates are from a mixed effects model with treatment, subject population, treatment by subject population interaction, baseline trough FEV1 and region as fixed effects and center nested within region as random effects. Full analysis set included all randomized subjects who received at least one dose of study drug.
Time Frame: baseline,12 weeks
Measure: Least Squares Mean (Standard Error); unit: liter
Arm/Group | QAW039 450 mg qd Non-atopic | Placebo Non-atopic | QAW039 450 mg qd Atopic | Fluticasone 150 µg Bid Atopic | Placebo Atopic
Number analyzed (Participants) | 91 | 93 | 50 | 41 | 52
liter | 0.05 (0.029) | 0.03 (0.029) | 0.06 (0.038) | 0.01 (0.042) | 0.05 (0.037)
Statistical Analysis 1: Comparison: QAW039 450 mg qd Non-atopic vs Placebo Non-atopic vs QAW039 450 mg qd Atopic vs Fluticasone 150 µg Bid Atopic vs Placebo Atopic; Test type: Superiority or Other; p = 0.9179, Mixed Models Analysis

4. Secondary Outcome: Change From Baseline in ACQ-6 Score at Week 12 Non-atopic and Atopic Patients at Week 12 - Full Analysis Set
Description: ACQ-6 consists of:5 items on symptoms, 1 item on rescue bronchodilator use, and 1 item on airway caliber (FEV1 % predicted). The ACQ was fully validated, including a minimal important difference (MID) or smallest change that could be considered clinically important (0.5). The ACQ was self-administered at the clinic and patients scored each item on a 7-point response scale: 0 = 'totally controlled' and 6 = 'severely uncontrolled.' Study staff scored question 7 based on % predicted FEV1 (ideally pre-bronchodilator). The total score=average of first 6 questions. Baseline=the ACQ-6 measurement taken prior to first dose of randomized study drug. The single missing score was interpolated by utilizing prior or subsequent completions of the questionnaire. Estimates were from a mixed effects model with treatment, subject population (non-atopic vs. atopic), treatment by subject population interaction, baseline ACQ-6 and region as fixed effects and center nested within region as random effects.
Time Frame: baseline,12 weeks
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | QAW039 450 mg qd Non-atopic | Placebo Non-atopic | QAW039 450 mg qd Atopic | Fluticasone 150 µg Bid Atopic | Placebo Atopic
Number analyzed (Participants) | 80 | 85 | 48 | 40 | 48
score | -0.05 (0.077) | -0.03 (0.073) | -0.25 (0.096) | -0.35 (0.104) | -0.18 (0.096)
Statistical Analysis 1: Comparison: QAW039 450 mg qd Non-atopic vs Placebo Non-atopic; Test type: Superiority or Other; least squares mean = -0.02, 95% CI 2-sided [-0.22 to 0.17], Standard Error of Mean 0.098
Statistical Analysis 2: Comparison: QAW039 450 mg qd Atopic vs Placebo Atopic; Test type: Superiority or Other; least sqares mean = -0.07, 95% CI 2-sided [-0.32 to 0.19], Standard Error of Mean 0.128
Statistical Analysis 3: Comparison: QAW039 450 mg qd Atopic vs Fluticasone 150 µg Bid Atopic; Test type: Superiority or Other; least squares mean = 0.10, 95% CI 2-sided [-0.16 to 0.37], Standard Error of Mean 0.134
Statistical Analysis 4: Comparison: Fluticasone 150 µg Bid Atopic vs Placebo Atopic; Test type: Superiority or Other; least squares mean = -0.17, 95% CI 2-sided [-0.43 to 0.09], Standard Error of Mean 0.134

5. Secondary Outcome: Change From Baseline in ACQ-6 Score at Week 12 Non-atopic Compared to Atopic Patients at Week 12 - Full Analysis Set
Description: as for outcome 4
Time Frame: baseline,12 weeks
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | QAW039 450 mg qd Non-atopic | Placebo Non-atopic | QAW039 450 mg qd Atopic | Fluticasone 150 µg Bid Atopic | Placebo Atopic
Number analyzed (Participants) | 80 | 85 | 48 | 40 | 48
score | -0.05 (0.077) | -0.03 (0.073) | -0.25 (0.096) | -0.35 (0.104) | -0.18 (0.096)
Statistical Analysis 1: Comparison: QAW039 450 mg qd Non-atopic vs Placebo Non-atopic vs QAW039 450 mg qd Atopic vs Fluticasone 150 µg Bid Atopic vs Placebo Atopic; Test type: Superiority or Other; p = 0.7930, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Timeframe for AE
Description: AE additional description
Groups:
- QAW039 450 mg qd: QAW039 450 mg qd
- Fluticasone 150 mcg Bid: Fluticasone 150 mcg bid
- Placebo: Placebo
Arm/Group | QAW039 450 mg qd | Fluticasone 150 mcg Bid | Placebo
Serious Adverse Events (participants affected / at risk) | 2/145 | 0/42 | 3/147
Other Adverse Events (participants affected / at risk) | 36/145 | 19/42 | 35/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 450 mg qd (N=145) | Fluticasone 150 mcg Bid (N=42) | Placebo (N=147)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0 | 0
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 1
OVARIAN CYST (Reproductive system and breast disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 450 mg qd (N=145) | Fluticasone 150 mcg Bid (N=42) | Placebo (N=147)
DENTAL CARIES (Gastrointestinal disorders) | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 1 | 1
ACUTE SINUSITIS (Infections and infestations) | 0 | 0 | 3
BRONCHITIS (Infections and infestations) | 3 | 0 | 4
CONJUNCTIVITIS VIRAL (Infections and infestations) | 0 | 1 | 0
INFLUENZA (Infections and infestations) | 2 | 0 | 3
NASOPHARYNGITIS (Infections and infestations) | 5 | 1 | 3
ORAL CANDIDIASIS (Infections and infestations) | 0 | 1 | 1
PHARYNGITIS (Infections and infestations) | 1 | 1 | 0
RHINITIS (Infections and infestations) | 2 | 2 | 0
SINUSITIS BACTERIAL (Infections and infestations) | 3 | 0 | 0
SKIN INFECTION (Infections and infestations) | 0 | 1 | 0
TONSILLITIS (Infections and infestations) | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 1 | 5
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1 | 3
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0
WOUND (Injury, poisoning and procedural complications) | 0 | 1 | 0
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1 | 1 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 | 2 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 3
SYNCOPE (Nervous system disorders) | 0 | 1 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 1 | 0
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 | 1 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 13
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.